CLINICAL TRIAL: NCT05667155
Title: Clinical Study of Cord Blood-derived CAR NK Cells Targeting CD19/CD70 in Refractory/Relapsed B-cell Non-Hodgkin Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-088
Record Dates: First submitted 2022-11-29; First posted 2022-12-28 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: B-cell Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CB dualCAR-NK19/70 (Experimental): All subjects were intravenously administrated with CB dualCAR-NK19/70
  Interventions: Biological: CB dualCAR-NK19/70

INTERVENTIONS:
Biological: CB dualCAR-NK19/70 — Lentiviral vector-transducted cord blood-derived NK cells to express anti-CD19/CD70 CAR and IL15

SUMMARY:
To study the safety and efficacy of cord blood-derived CAR-NK cells targeting CD19/CD70 in patients with B-cell non-Hodgkin's lymphoma

DETAILED DESCRIPTION:
This is a single-center, open, one-arm, dose-escalation study to observe the safety and efficacy of cord blood-derived dualCAR-NK19/70 cells in patients with B-cell non-Hodgkin lymphoma.9-18 patients are planned to be enrolled in the dose-escalation trial (2×10^6 cells/kg, 4×10^6 cells/kg, 8×10^6 cells/kg) . Each dose was given once a week for 3 weeks.The primary endpoints are DLT, MTD, and the second endpionts are the overall response rates (CR and PR), overall survival, and progression-free survival. Based on the results in the dose-escalation trial, the recommended dose will be determined. Another 30 patients will be enrolled to estimate the safety and efficacy of CB CAR-NK019 under the best dose.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in the study and sign the informed consent;
2. Age 18-75, male and female;
3. Histologically confirmed diffuse large B-cell lymphoma (DLBCL), transformed follicular lymphoma (tFL), primary mediastinal B-cell lymphoma (PMBCL), mantle cell lymphoma (MCL), and other inert B-cell NHL transforming types:

(1)refractory or recurrent DLBCL and tFL must be approved by 2 line immune disease relapse after chemotherapy treatment; (2) refractory definition large B cell lymphoma (research SCHOLAR - 1 standard) : more than 4 courses first-line immune chemotherapy disease progression; The stable time of the disease is equal to or less than 6 months; Or disease progression or recurrence within 12 months after autologous hematopoietic stem cell transplantation; (3) refractory or recurrent MCL must be 1 line with immune chemotherapy; BTK inhibitors are resistant or intolerant as 2-line therapy; (4)always treatment must include CD20 single resistance (unless the subjects for CD20 negative) and anthracycline-based;

4. There was at least one measurable lesion with the longest diameter ≥1.5 cm;

5. Predicted survival ≥12 weeks;

6. The expression of CD19 or CD70 in biopsy sections of tumor tissue was positive;

7. ECOG score 0-2;

8. Adequate reserve of organ functions:

1. cereal third transaminase, aspartate aminotransferase 2.5 x or less UNL (upper limit of normal);
2. creatinine clearance (Cockcroft - Gault method) or 60 mL/min.
3. serum total bilirubin and alkaline phosphatase (1.5 x or less UNL.
4. glomerular filtration rate > 50 mL/min
5. heart ejection fraction (EF) 45% or higher;
6. indoor natural air environment, basic oxygen saturation > 92%
7. blood routine: neutrophils absolute number > 1000 cells/mm3, platelet count 45 x109, 8.0 g/dL hemoglobin;

9. Allowed to have received a previous stem cell transplant

10. Approved anti-B-cell lymphoma therapies, such as systemic chemotherapy, systemic radiotherapy and immunotherapy, had been completed for at least 3 weeks before the study. The eluting period of targeted drug regimens without chemotherapy was 2 weeks;

11. Patients who had previously received CAR T cell therapy and failed to respond to a 3-month evaluation or relapsed were admitted;

12. Female subjects of childbearing age must test negative for pregnancy and agree to use effective contraceptive methods during the trial

13. Two tests have come back negative for COVID-19.

Exclusion Criteria:

1. Allergic to any of the components of cell products;
2. History of other tumors;
3. Acute GvHD or generalized chronic GvHD with grade II-IV (Glucksberg standard) after previous allogeneic hematopoietic stem cell transplantation; Or being treated with anti-GVHD;
4. Had received gene therapy in the past 3 months;
5. Active infections requiring treatment (other than simple urinary tract infections and bacterial pharyngitis), however, prophylactic antibiotics, antiviral and antifungal infections are allowed;
6. Subjects infected with hepatitis B (HBsAg positive, but HBV-DNA<103 is not excluded) or hepatitis C virus (including virus carriers), syphilis and other acquired and congenital immunodeficiency diseases, including but not limited to HIV-infected persons;
7. Subjects with Grade III or IV cardiac insufficiency according to the New York Heart Association Cardiac Function Grading criteria;
8. Patients who received antitumor therapy in the early stage but the toxicity reaction did not recover (CTCAE 5.0 toxicity reaction did not recover to ≤ level 1, except fatigue, anorexia and alopecia);
9. Subjects with a history of epilepsy or other central nervous system diseases;
10. Skull enhanced CT or MRI showing evidence of central nervous system lymphoma;
11. Lactating women who refuse to stop breastfeeding;
12. Any other circumstances that the investigator believes may increase the subject's risk or interfere with the test results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLTs) | Up to 28 days
  To evaluate the safety, tolerability, and determine the recommended dosage of cord blood-derived Anti-CD19 CAR-NK Cell Therapy for B-cell Non-Hodgkin Lymphoma

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 2 years
  To determine the anti-tumor effectivity of CB dualCAR-NK19/70
Overall response rate (ORR) | Up to 2 years
  To determine the anti-tumor effectivity of CB dualCAR-NK19/70
Duration of response (DOR) | Up to 2 years
  To determine the anti-tumor effectivity of CB dualCAR-NK19/70
Complete response rate (CR) | Up to 2 years
  To determine the anti-tumor effectivity of CB dualCAR-NK19/70
Partial response rate (PR) | Up to 2 years
  To determine the anti-tumor effectivity of CB dualCAR-NK19/70
Progression free survival (PFS) | Up to 2 years
  To determine the anti-tumor effectivity of CB dualCAR-NK19/70

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Wenbin, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No